CLINICAL TRIAL: NCT06348849
Title: The Desensitising Effect of Nanosilver Fluoride Compared to Low-Level Laser Therapy in Molar-Incisor Hypomineralisation: A Randomised Controlled Clinical Trial
Brief Title: The Desensitising Effect of Nanosilver Fluoride in Molar-Incisor Hypomineralisation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Nouran Nabil, Instructor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0797-11/2023
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Molar Incisor Hypomineralization; Hypersensitivity
Keywords: Nanosilver fluoride; Low-level laser therapy; Desensitising; Molar-incisor hypomineralisation; First permanent molars; Pediatric; Clinical trial; Nanosilver; LLLT
MeSH Terms: conditions — Molar Hypomineralization; Hypersensitivity | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-level laser therapy (Active Comparator): These hypersensitive molars with MIH will receive low-level laser therapy.
  Interventions: Device: Low-level laser therapy
- Nanosilver fluoride (Experimental): These hypersensitive molars with MIH will receive nanosilver fluoride treatment.
  Interventions: Drug: Nanosilver fluoride

INTERVENTIONS:
Device: Low-level laser therapy — Wavelength 980nm (SmartM, Lasotronix, Poland)
  Arms: Low-level laser therapy
Drug: Nanosilver fluoride — Optimized synthesis of Nanosilver Fluoride
  Arms: Nanosilver fluoride

SUMMARY:
The aim of the current study is to assess the desensitising effect of nanosilver fluoride on first permanent molars (FPMs) in patients with MIH in comparison to low-level laser therapy.

ELIGIBILITY:
Inclusion Criteria:

* The presence of at least one hypersensitive first permanent molar in MIH patient (using the Schiff Cold Air Sensitivity Scale (SCASS)).
* Completion of an informed consent to participate in the study.

Exclusion Criteria:

* Hypomineralised molars resulting from other medical conditions, such as enamel malformations associated with syndromes, dental fluorosis, enamel hypoplasia, amelogenesis imperfecta, and dental caries.
* The presence of active tooth decay or defective restorations in the tooth under examination which can confound the aetiology of hypersensitivity with pulpitis.
* The presence of pulpal symptoms.
* Having undergone any professional desensitising treatment in the previous 6 months.
* Having used a desensitising paste other than habitual toothpaste in the previous 3 months.
* Use of anti-inflammatory drugs or analgesics at the time of recruitment.
* Allergy or sensitivity to silver or any of the materials included in the study.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Desensitising effect in hypersensitive MIH molars | 1 month
  This will be performed using Schiff Cold Air Sensitivity Scale (SCASS). The SCASS will be used to assess subject response to this stimulus (0=no response to the stimulus; 1=no response to the stimulus, patient considers stimulus to be painful; 2= response to stimulus, patient moves from the stimulus; 3= response to the stimulus, patient moves from the stimulus and requests immediate discontinuation of the stimulus)

SECONDARY OUTCOMES:
Change in the plaque index scores | 1 month
  This will be assessed using the modified plaque index (PlI) of Silness and Löe. Each tooth will be scored from 0 (lowest) to 3 (highest) according to the amount of plaque accumulation. The total score will be determined by calculating the average score of the examined teeth.
Change in children's frequency of toothbrushing | 1 month
  The frequency of toothbrushing will be assessed using a question adapted from the World Health Organization (WHO) questionnaire- child version. The parent will be asked about the number of times his/her child brushes their teeth (never - several times a month - once a week - several times a week - once daily - twice or more daily)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nabil N, Sharaf AA, Essawy MM, Soliman RS. The Desensitizing Effect of Nanosilver Fluoride Compared to Photobiomodulation Therapy in Molar-Incisor Hypomineralization: A Randomized Clinical Trial. J Evid Based Dent Pract. 2025 Sep;25(3):102139. doi: 10.1016/j.jebdp.2025.102139. Epub 2025 Mar 14. PMID 40716831